CLINICAL TRIAL: NCT00290888
Title: Arthroscopic Rotator Cuff Repair With and Without Arthroscopic Acromioplasty in the Treatment of Full Thickness Rotator Cuff
Brief Title: Arthroscopic Rotator Cuff Repair of Full Thickness Tears With and Without Arthroscopic Acromioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panam Clinic (Other)
Responsible Party: Principal Investigator, Peter MacDonald, Department Head, Orthopaedics, Panam Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2004:045
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Rotator Cuff Tear; Shoulder Impingement Syndrome
Keywords: Rotator Cuff Tear; Tendon Repair; Acromioplasty; Arthroscopy; Orthopedic Surgery
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACR (Active Comparator): Arthroscopic rotator cuff repair without acromioplasty
  Interventions: Procedure: Acromioplasty
- ACR-A (Experimental): Arthorscopic rotator cuff repair with acromioplasty
  Interventions: Procedure: Acromioplasty

INTERVENTIONS:
Procedure: Acromioplasty

SUMMARY:
Surgical repair of full thickness tears of the rotator cuff is a controversial issue, with several procedures currently being used to treat the tear. The two most common treatments at this point in time are arthroscopic cuff repair with and without acromioplasty. However, an arthroscopic cuff repair without acromioplasty may offer the same degree of improvement as one that includes acromioplasty, but without threatening the shoulder stability that is provided by the acromion and coracoacromial ligament. This prospective study examines the hypothesis that appropriate shoulder function can be restored through the execution of the traditional arthroscopic cuff repair without acromioplasty.

DETAILED DESCRIPTION:
There exists some controversy in the current trend in repair of full thickness tears of the rotator cuff. The two most common treatments at this point in time are arthroscopic cuff repair with and without acromioplasty. The purpose of acromioplasty is to create adequate space for the rotator cuff tendons. Arthroscopic acromioplasty involves the removal of the subacromial bursa, resection of the coracoacromial ligament and anteroinferior portion of the acromion, and resection of any osteophytes from the acromioclavicular joint that are thought to be contributing to impingement. However, acromioplasty without cuff repair has been reported to have both good and poor results, showing that the technique may be suspect in repair of full thickness tears alone.

The purpose of this study is to compare the effectiveness of arthroscopic cuff repair with acromioplasty to arthroscopic cuff repair without acromioplasty in repair of full thickness tears of the rotator cuff.

We hypothesize that there will be a significant clinical improvement in quality of life in patients who receive a rotator cuff repair without acromioplasty compared to those who receive a cuff repair with acromioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older
* Complete rotator cuff tear up to 4 cm in size
* Persistent pain and functional disability for at least 6 months
* Failure of conservative treatment
* Establishment of final eligibility based upon visual exam of rotator cuff tear during surgery and determination of repairability

Exclusion Criteria:

* Evidence of significant osteoarthritis or cartilage damage in the shoulder
* Evidence of glenohumeral instability including Bankart lesions and labral tears of any type
* Previous surgeries of the shoulder
* Evidence of major joint trauma, infection, or necrosis in the shoulder
* Patients with partial thickness tears of the rotator cuff
* Patients unable to provide informed consent due to language barrier or mental status
* Patients with a major medical condition that would affect quality of life and influence the results of the study
* Patients with worker compensation claims
* Patients unwilling to be followed for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter MacDonald, MD, FRCS(C), Principal Investigator — Panam Clinic Orthopedics and Sports Medicine/University of Manitoba
Locations (1):
- Panam Clinic, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Kirkley A, Griffin S, McLintock H, Ng L. The development and evaluation of a disease-specific quality of life measurement tool for shoulder instability. The Western Ontario Shoulder Instability Index (WOSI). Am J Sports Med. 1998 Nov-Dec;26(6):764-72. doi: 10.1177/03635465980260060501. PMID 9850776
- [Background] Baker CL, Liu SH. Comparison of open and arthroscopically assisted rotator cuff repairs. Am J Sports Med. 1995 Jan-Feb;23(1):99-104. doi: 10.1177/036354659502300117. PMID 7726359
- [Background] Gartsman GM. Arthroscopic assessment of rotator cuff tear reparability. Arthroscopy. 1996 Oct;12(5):546-9. doi: 10.1016/s0749-8063(96)90192-9. PMID 8902127
- [Background] Miller C, Savoie FH. Glenohumeral abnormalities associated with full-thickness tears of the rotator cuff. Orthop Rev. 1994 Feb;23(2):159-62. PMID 8196974
- [Background] Budoff JE, Nirschl RP, Guidi EJ. Debridement of partial-thickness tears of the rotator cuff without acromioplasty. Long-term follow-up and review of the literature. J Bone Joint Surg Am. 1998 May;80(5):733-48. doi: 10.2106/00004623-199805000-00016. No abstract available. PMID 9611036
- [Background] Gartsman GM, Taverna E. The incidence of glenohumeral joint abnormalities associated with full-thickness, reparable rotator cuff tears. Arthroscopy. 1997 Aug;13(4):450-5. doi: 10.1016/s0749-8063(97)90123-7. PMID 9276051
- [Background] Esch JC. Arthroscopic subacromial decompression and postoperative management. Orthop Clin North Am. 1993 Jan;24(1):161-71. PMID 8421609
- [Background] Levy HJ, Gardner RD, Lemak LJ. Arthroscopic subacromial decompression in the treatment of full-thickness rotator cuff tears. Arthroscopy. 1991;7(1):8-13. doi: 10.1016/0749-8063(91)90071-5. PMID 2009126
- [Background] Cofield RH. Rotator cuff disease of the shoulder. J Bone Joint Surg Am. 1985 Jul;67(6):974-9. No abstract available. PMID 4019548
- [Background] Bokor DJ, Hawkins RJ, Huckell GH, Angelo RL, Schickendantz MS. Results of nonoperative management of full-thickness tears of the rotator cuff. Clin Orthop Relat Res. 1993 Sep;(294):103-10. PMID 8358901
- [Background] Ellman H, Kay SP, Wirth M. Arthroscopic treatment of full-thickness rotator cuff tears: 2- to 7-year follow-up study. Arthroscopy. 1993;9(2):195-200. doi: 10.1016/s0749-8063(05)80374-3. PMID 8461081
- [Background] Neer CS 2nd. Anterior acromioplasty for the chronic impingement syndrome in the shoulder: a preliminary report. J Bone Joint Surg Am. 1972 Jan;54(1):41-50. No abstract available. PMID 5054450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 86 patients were randomized to either ACR-A or ACR
Groups:
- Arthroscopic Rotator Cuff Repair Without Acromioplasty: ACR
  Acromioplasty
- Arthorscopic Rotator Cuff Repair With Acromioplasty: ACR-A
  Acromioplasty
Period: Overall Study
Arm/Group | Arthroscopic Rotator Cuff Repair Without Acromioplasty | Arthorscopic Rotator Cuff Repair With Acromioplasty
Started | 41 | 45
Completed | 38 | 44
Not Completed | 3 | 1
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arthroscopic Rotator Cuff Repair Without Acromioplasty: Arthroscopic rotator cuff repair without acromioplasty (ACR)
- Arthroscopic Rotator Cuff Repair With Acromioplasty: Arthroscopic rotator cuff repair with acromioplasty (ACR-A)
- Total: Total of all reporting groups
Arm/Group | Arthroscopic Rotator Cuff Repair Without Acromioplasty | Arthroscopic Rotator Cuff Repair With Acromioplasty | Total
Number analyzed (Participants) | 41 | 45 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (9.5) | 56.2 (7.9) | 56.7 (8.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 45 | 86
  >=65 years | 0 | 0 | 0
Gender [Number; unit: participants]
  Female | 15 | 14 | 29
  Male | 30 | 24 | 54
Region of Enrollment [Number; unit: participants]
  Canada | 41 | 45 | 86

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario Rotator Cuff Index (WORC)
Description: Calculated as percentage with an increase in score indicating an improvement in outcome.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: percentage of total score
Groups:
- Arthroscopic Rotator Cuff Repair Without Acromioplasty: ACR
- Arthroscopic Rotator Cuff Repair With Acromioplasty: ACR-A
  Acromioplasty
Arm/Group | Arthroscopic Rotator Cuff Repair Without Acromioplasty | Arthroscopic Rotator Cuff Repair With Acromioplasty
Number analyzed (Participants) | 38 | 44
percentage of total score | 80.5 (22.3) | 86.7 (16.2)

2. Primary Outcome: American Shoulder and Elbow Surgeons Standardized Form for the Assessment of the Shoulder (ASES)
Description: Calculated as a percentage with an increase in score reflecting an improvement in outcome.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: percentage of total score
Arm/Group | Arthroscopic Rotator Cuff Repair Without Acromioplasty | Arthorscopic Rotator Cuff Repair With Acromioplasty
Number analyzed (Participants) | 38 | 44
percentage of total score | 84.6 (20.1) | 89.8 (14.4)

3. Secondary Outcome: Shoulder Range of Motion
Time Frame: 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Upper Extremity Strength Grading
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Arthroscopic Rotator Cuff Repair Without Acromioplasty | Arthroscopic Rotator Cuff Repair With Acromioplasty
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/45
Other Adverse Events (participants affected / at risk) | 0/41 | 0/45

LIMITATIONS AND CAVEATS:
Variation in surgical technique and post-op rehabilitation. We do not have confirmation of cuff healing status as no imaging was carried out post-operatively. Assessment of AC morphology is subjective & based solely on pre-operative radiographs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes